CLINICAL TRIAL: NCT03088020
Title: International Congenital Central Hypoventilation Syndrome (CCHS) REDCap Registry and CCHS Secure Health-hub Advancing Research Efforts
Brief Title: International Congenital Central Hypoventilation Syndrome (CCHS) Registry and CCHS SHARE
Status: Recruiting | Type: Observational
Sponsor: Debra Weese-Mayer (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other); The Chicago Community Trust (Other)
Responsible Party: Sponsor-Investigator, Debra Weese-Mayer, Professor of Pediatric Autonomic Medicine, Northwestern University Feinberg School of Medicine; Chief, Center for Autonomic Medicine in Pediatrics (CAMP), Ann & Robert H. Lurie Children's Hospital and Stanley Manne Children's Research Institute, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Other Study IDs: 2013-15203
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Congenital Central Hypoventilation Syndrome
Keywords: CCHS; PHOX2B; Paired-like Homeobox gene PHOX2B; autonomic nervous system dysregulation; control of breathing; Hirschsprung disease; neural crest tumors; neuroblastoma; ganglioneuroma; ganglioneuroblastoma; artificial ventilation; diaphragm pacing
MeSH Terms: conditions — Congenital central hypoventilation syndrome; Hirschsprung Disease; Neuroblastoma; Ganglioneuroma; Ganglioneuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Center for Autonomic Medicine in Pediatrics (CAMP), in collaboration with leading CCHS clinicians, scientists, and patient advocacy groups around the world has built the first International CCHS (Congenital Central Hypoventilation Syndrome REDCap (Research Electronic Data Capture) Registry. This registry is an international collaboration to capture CCHS natural history data with CCHS patients and their physicians recruited from around the world. This registry is part of a CCHS natural history study that includes the CCHS Secure Health-hub Advancing Research Efforts (CCHS-SHARE), a natural history data platform shared with the broader CCHS research and patient community to house extensive longitudinal, de-identified data. Inclusion of registry data in CCHS-SHARE is optional.

The purpose of this IRB-approved research study is to gain a better understanding of the natural history of CCHS, including the various clinical manifestations of CCHS with advancing age, and as related to each patient's specific PHOX2B mutation. With a better understanding of CCHS natural history, we will be able to better anticipate healthcare needs and to provide more accurate guidelines to healthcare providers world-wide in caring for patients with CCHS.

The study aims to obtain detailed phenotypic information (information about health and well-being) on patients with CCHS and their families. Participation would require filling out a confidential survey that asks questions regarding phenotype and past medical history. Involvement in the project is completely voluntary and there is no compensation for taking part. However, this project will help us learn more about this disease, with the goal of advancing treatment.

DETAILED DESCRIPTION:
CCHS is a disorder characterized by alveolar hypoventilation with a control of breathing deficit, and symptoms of autonomic nervous system (ANS) dysregulation (ANSD). This study aims to develop a patient registry for CCHS, which will provide crucial insight into disease development, improving outcome in these children through improving early recognition of the disorder, understanding the phenotypic spectrum, and evolution of CCHS natural history. Data will be stored in REDCap (Research Electronic Data Capture) system a secure web application designed exclusively to support data capture for research studies in a secure manner. The REDCap server is hosted securely at Northwestern University, behind a firewall, with virus protection, and using Secure Socket Layer (SSL) authentication to encrypt communication between a user and the server. Protected Health Information (PHI) will be labeled as such in the database and access to it will be restricted to the Principal Investigator (PI) and key personnel participating in the consent process and follow up contact of participants.

Participants in the International CCHS REDCap Registry will be identified and recruited from CAMP's registry of new, current, and past CCHS referrals, including CCHS patients referred for PHOX2B testing and/or consultation. Additionally, patients may also be recruited via the internet using emails, Facebook pages, and mailing lists for family groups. Anyone interested will be offered inclusion into the International CCHS Registry. Participants will be able to participate remotely, from their homes or locations where they have internet, phone, and computer access.

Data collected through the REDCap registry will be de-identified and analyzed. Patients enrolled in this study will be offered participation in CCHS-SHARE and the NIH Global Rare Disease Registry (GRDR). These are both optional parts of the study, and are not required for inclusion. The CCHS-SHARE is a data repository that houses de-identified clinical and registry data on CCHS patients, empowering data sharing across the CCHS research community. The GRDR is established by the NIH Office of Rare Disease Research. The goal of the GRDR is to establish a data repository of de-identified patient data, aggregated in a standardized manner, using Common Data Elements (CDEs) and standardized terminology. De-identification of patient's data will utilize the Global Unique Identifiers (GUID) system. Lurie Children's Hospital will retain ownership of all data shared with CCHS-SHARE and the GRDR. The de-identified data in CCHS-SHARE and GRDR will be available to all investigators to enable analyses across many rare diseases and to facilitate various biomedical studies, including clinical trials, in pursuit of developing drugs and therapeutics to improve the healthcare and the quality of life for the many millions of people who are diagnosed with rare diseases.

Any patient agreeing to be part of CCHS-SHARE and/or GRDR will have their data de-identified and this de-identified data exported and shared with CCHS-SHARE and the GRDR. These participants are also given the option to be contacted for participation in clinical trials. If this option is chosen, any researcher accessing de-identified information through CCHS-SHARE and GRDR and planning to conduct a clinical trial will be allowed to contact the CAMP project coordinator to ask that patients fitting the profile of needed participants be contacted and offered inclusion. No de-identified information will be shared with researchers outside of CAMP, rather the CAMP project coordinator will contact identified patients fitting participation criteria to share contact information and details for the clinical trial. Interested patients will then be given to the option to contact researchers conducting clinical trials at their discretion.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with PHOX2B mutation-confirmed CCHS.

Exclusion Criteria:

* Individuals without PHOX2B mutation-confirmed CCHS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CCHS patients with confirmed PHOX2B mutations
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-06-24 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal phenotype in CCHS | 20 years
  Collection of longitudinal disease history in 400 CCHS patients

SECONDARY OUTCOMES:
Sensitive markers of disease progression by PHOX2B mutation/genotype | 20 years
  Evaluate patient reported outcome measures to determine sensitive markers of disease progression for use in intervention trials
Integration of CCHS Registry and Global Rare Diseases Patient Registry (GRDR) | 20 years
  Develop a patient registry for CCHS for use with the CCHS Secure Health-hub Advancing Research Efforts" (CCHS-SHARE) and the global rare diseases patient registry and data repository (GRDR)

CONTACTS AND LOCATIONS:
Overall Officials: Debra E Weese-Mayer, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago and the Stanley Manne Children's Research Institute, Chicago, Illinois, United States

REFERENCES:
- See also: CAMP Website about International CCHS REDCap Registry — https://www.luriechildrens.org/en/specialties-conditions/autonomic-medicine/research/